CLINICAL TRIAL: NCT02948322
Title: Cardiac Structure and Function in Acromegalic Patients: A Cardiac Magnetic Resonance Imaging Study
Brief Title: Cardiac (CMRI) Assessment of Acromegaly
Acronym: ACROCOEUR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: P121004
Record Dates: First submitted 2015-12-08; First posted 2016-10-28 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2016-10

CONDITIONS: Acromegaly
Keywords: Acromegaly,; water retention; myocardial fibrosis; left ventricular hypertrophy; left ventricular dysfunction
MeSH Terms: conditions — Acromegaly; Hypertrophy, Left Ventricular; Ventricular Dysfunction, Left | interventions — Gadolinium; Glucose Tolerance Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OGTT, CMRI with gadolinium in patients (Experimental): Patients with acromegaly will be investigated
  Interventions: Device: CMRI; Drug: Gadolinium; Procedure: OGTT
- OGTT, CMRI with gadolinium in volunteers (Active Comparator): Age-, sex- and BMI-matched healthy volunteers will be investigated
  Interventions: Device: CMRI; Drug: Gadolinium; Procedure: OGTT

INTERVENTIONS:
Device: CMRI — Myocardial Imaging (CMRI) will be performed in patients (at baseline and 6 month after treatment) and healthy volunteers (baseline)
Drug: Gadolinium — gadolinium injection will be performed during CMRI in patients and healthy volunteers.
  Other Names: Gadolinium injection
Procedure: OGTT — Growth Hormon (GH) secretion and metabolic status of the acromegalic will be evaluated by an measure of plasma glucose, insulin and GH (OGTT), and insulin-like growth factor-1 (IGF-I) will be measured in patients and healthy volunteers.

SUMMARY:
In this study, the investigators will evaluate the cardiac structure and function, focusing on the myocardial water content and interstitial fibrosis, in patients with active acromegaly in comparison with 1) healthy volunteers, 2) the same acromegalic patients that have received efficient therapy.

The investigators hypothesize that the myocardial water content in acromegaly is increased as these patients present with sodium and water retention and that this myocardial water infiltration will improve with efficient treatment of the disease. They will thus assess using CMRI, this parameter by measuring the myocardial transverse relaxation time (T2), reflecting water content in the myocardium.

DETAILED DESCRIPTION:
Patients with acromegaly have left ventricular (LV) hypertrophy and dysfunction on echocardiography, but only very few studies have been performed using cardiac magnetic resonance imaging (CMRI), currently the reference modality is assessment in cardiac geometry function. In addition, no data are available on right ventricular (RV) and atrial structure and function. The pathophysiology of the cardiac involvement in acromegaly may be related to increase myocardiac water content and/or interstitial myocardiac fibrosis.

The main objective of sthe study is to compare the myocardial water content in patients with acromegaly and in healthy volunteers. Secondary objectives of the study are to evaluate :

1. interstitial fibrosis and the structure and the function of LV and RV in acromegalic patients in comparison with healthy volunteers;
2. the reversibility of the cardiac involvement (water content, fibrosis, LV and RV structure and function) after efficient treatment of acromegaly;
3. the elasticity of aorta in acromegalic patients in comparison with healthy volunteers and with the post-treatment state. Twenty acromegalic patients will be included in order to dispose of 15 patients that will completed the study and the same number of age- and BMI-adjusted healthy volunteers will be included.

ELIGIBILITY:
Inclusion Criteria:

* Active acromegaly as defined by the usual diagnostic criteria (de novo patients or patients uncontrolled by previous treatments).
* Healthy volunteers matched for age, sex and BMI with the patients of the group 1

Exclusion Criteria:

* History of coronary heart disease (acute or chronic myocardial ischemia)
* Acute or chronic renal failure (creatinin clearance 30 mL/min/l,73m2)
* Contraindication of MRI
* Hypersensitivity to gadolinium
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-12; Primary Completion 2017-06-09 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Myocardial transverse relaxation time (T2), reflecting water content assessed by CMRI | Baseline in acromegalic patients; at the 1 day evaluation visit in healthy volunteers
  This outcome will be compared between patients and healthy volunteers.
Change from baseline Myocardial transverse relaxation time (T2) at 6 months, reflecting water content assessed by CMRI | Baseline and 6 months after beginning of the treatment in acromegalic patients

SECONDARY OUTCOMES:
Dense myocardial fibrosis | Baseline in acromegalic patients; at the 1 day evaluation visit in healthy volunteers
  The dense myocardial fibrosis will be depicted by late gadolinium enhancement.
Interstitial myocardial fibrosis | Baseline in acromegalic patients; at the 1 day evaluation visit in healthy volunteers
  Interstitial myocardial fibrosis will be quantified by T1 measurements before and after gadolinium injection.
Cardiac morphology will also be assessed CMRI | Baseline in acromegalic patients; at the 1 day evaluation visit in healthy volunteers
Function including Left Ventricular mass index will also be assessed CMRI | Baseline in acromegalic patients; at the 1 day evaluation visit in healthy volunteers
Function including Left Auricular ejection fractions will also be assessed CMRI | Baseline in acromegalic patients; at the 1 day evaluation visit in healthy volunteers
Function including Left Ventricular ejection fractions will also be assessed CMRI | Baseline in acromegalic patients; at the 1 day evaluation visit in healthy volunteers
Function including Right Ventricular ejection fractions will also be assessed CMRI | Baseline in acromegalic patients; at the 1 day evaluation visit in healthy volunteers
Function including Left Ventricular and Right Ventricular stroke volumes will also be assessed CMRI | Baseline in acromegalic patients; at the 1 day evaluation visit in healthy volunteers
Change from baseline Dense myocardial fibrosis at 6 months | Baseline and 6 months after beginning of the treatment in acromegalic patients
  "The dense myocardial fibrosis will be depicted by late gadolinium enhancement.
Change from baseline interstitial myocardial fibrosis at 6 months | Baseline and 6 months after beginning of the treatment in acromegalic patients

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CHANSON, MD, PhDI, Principal Investigator — AP-HP, Bicêtre Hospital
Locations (1):
- AP-HP, Bicêtre Hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wolf P, Bouazizi K, Kachenoura N, Piedvache C, Gallo A, Salenave S, Maione L, Young J, Prigent M, Lecoq AL, Kuhn E, Agostini H, Trabado S, Redheuil A, Chanson P, Kamenicky P. Increase in intracellular and extracellular myocardial mass in patients with acromegaly: a cardiac magnetic resonance imaging study. Eur J Endocrinol. 2023 Aug 2;189(2):199-207. doi: 10.1093/ejendo/lvad105. PMID 37549351